CLINICAL TRIAL: NCT03105570
Title: The Oncological Safety and Cosmetic Outcome of Areola Sparing Mastectomy : a Single Arm, Prospective, Cohort Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Houpu Yang, Principal Investigator, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASM-China
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Breast Neoplasms
Keywords: breast neoplasms; Mastectomy, Subcutaneous; Areola
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Armed, prospective, open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Areola sparing mastectomy. (Experimental): Eligible patients undergo areola sparing mastectomy.
  Interventions: Procedure: Areola Sparing Mastectomy

INTERVENTIONS:
Procedure: Areola Sparing Mastectomy — A small circular incision would be made to separate nipple from breast and an additional incision directly extended from nipple or located at other part of breast such as infra-mammary fold and subaxillary area would be made to remove the total mammary parenchyma. Routine implant based or flap base reconstruction would be performed subsequentially. Nipple reconstruction is optional.
  Other Names: Nipple coring

SUMMARY:
To balance the oncological safety and cosmetic outcome is the basic principle of modern breast surgery. To preserve the nipple-areolar complex shows attractive cosmetic advantage but concerns regarding local recurrence make the oncological safety of nipple sparing mastectomy a controversial issue. Since the involvement of areolar pigmented skin by cancer is rare compared to that of nipple, we designed the current study to investigate the oncological safety and cosmetic outcome of Areola Sparing Mastectomy.

DETAILED DESCRIPTION:
Primary breast cancer originated from areolae is rare. We hypothesized that nipple and areola are two separate anatomy tissue and have different oncological impact on the treatment of breast cancer. Areola Sparing Mastectomy (ASM) is a innovative procedure that involves of removal of nipple and preservation of areola the pigmented skin of which would improve the cosmetic outcome of mastectomy and lead to a illusion of congenital crater nipple in some patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive or in situ breast cancer.
* cTis-2N0-1M0.
* Indicated for total mastectomy and desire immediate breast reconstruction.

Exclusion Criteria:

* cT3-4 or cN2-N3 breast cancer.
* Retraction of nipple or areola.
* Involvement of subcutaneous layer by cancer on ultrasound or MRI.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of areolar area | Five years after initial surgery
  The frequency of histologically confirmed recurrence on the preserved pigmented areolar area.

SECONDARY OUTCOMES:
Cosmetic effect of reconstructed breast | 2-4 weeks after surgery; 2 years and 5 years after surgery.
  The cosmetic results evaluated by a surgeon and a nurse through reviewing photographs.
Adverse effect of surgery | 4 weeks after surgery.
  Wound dehiscence, infection, suture exposure and extrusion.
Disease free survival | 5 year after surgery
  Survival time to any recurrence and any cause death.

CONTACTS AND LOCATIONS:
Overall Officials: Shu Wang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No